CLINICAL TRIAL: NCT03805464
Title: Characterizing Changes in Knee Joint Loading With Wearable Sensor Technology Following an Experimental Knee Joint Effusion
Brief Title: Walking Gait Biomechanics Following Knee Joint Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00100862
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-02

CONDITIONS: Knee Injuries; Knee Osteoarthritis
Keywords: biomechanics; inertial measurement unit
MeSH Terms: conditions — Knee Injuries; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Knee Joint Effusion (Experimental): Participants will receive a one-time injection of 60mL of sterile saline into the suprapatellar space of the dominant lower extremity. This injection will be conducted under ultrasound guidance by a board-certified orthopedic surgeon.
  Interventions: Other: Knee Joint Effusion

INTERVENTIONS:
Other: Knee Joint Effusion — 60mL saline injection into the supra-patellar region of the knee

SUMMARY:
The purpose of this study is to determine the sensitivity of a wearable sensor to detect changes in knee joint loading using an experimental knee joint effusion as a model for a common clinical physiological alteration in joint status. The rationale for this project is that it will establish the efficacy of an inexpensive, clinically, and publicly available device that can detect changes in biomechanical loading due to acute physiologic change in joint status. The study will utilize a cross-sectional cohort study design and will seek to enroll 25 male and female healthy adult participants (18-35 yo). Participants will report to the laboratory for three total sessions (Session 1: informed consent and task familiarization; Session 2: testing; Session 3: knee joint status assessment). The primary outcomes of interest include lower extremity thigh and shank acceleration and velocity data (wearable sensor data), lower extermity 3D kinematics and kinetics (motion capture data), and lower extremity muscle function (EMG data) during walking gait, as well as functional balance and patient-reported subjective outcomes. Data will be analyzed by calculating change scores from the pre- to post-experimental effusion outcome measure testing. Paired-samples t-tests and Cohen's d effect sizes will be used to assess changed in wearable sensor data from pre- to post-experimental effusion. Correlation statistics will be used to determine if there are association between the motion capture and wearable sensor data. The potential risks associated with an experimental joint effusion will be addressed by maintaining appropriate sterile conditions and having the participant check-in with the PI (licensed healthcare provider) at 48 hours following testing session.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Chronological age 18-35 at the time of study participation
* Physically active (at least 30 minutes of physical activity, 3x/week)
* Tegner Activity Scale score at least 5/10

Exclusion Criteria:

* History of lower extremity or lumbar spine surgery.
* History of lower extremity or lumbar spine injury in the prior 6 months.
* History of major ligamentous damage.
* Current knee pain.
* Known neurological condition, autoimmune condition, cardiovascular disease.
* History of epilepsy, seizures, concussion within the prior 6 months.
* Currently taking pain altering medication.
* Fear of needles
* Unable to read and understand English language
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Change in Peak Vertical Ground Reaction Force | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Kinetic Loading Variable
Change in Peak Internal Knee Extension Moment | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Kinetic Loading Variable
Change in Peak Knee Power | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Kinetic Loading Variable
Change in Shank Acceleration | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Accelerometer Variable
Change in Thigh Acceleration | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Accelerometer Variable
Change in Shank Angular Velocity | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Gyroscope Variable
Change in Thigh Angular Velocity | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Gyroscope Variable

SECONDARY OUTCOMES:
Change in Quadriceps EMG | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Muscle Activity Variable
Change in Hamstring EMG | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Muscle Activity Variable
Change in Visual Analog Scale Pain | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Pain Variable
Change in International Knee Documentation Committee | Immediately Pre- (10 minutes) and Post- (10 minutes) Effusion
  Self-Reported Disability Variable

CONTACTS AND LOCATIONS:
Locations (1):
- Michael W. Krzyzewski Human Performance Laboratory, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No